CLINICAL TRIAL: NCT03416049
Title: A Sham Controlled Study to Compare the Effectiveness of Three Different Power Levels of PEMF Devices in the Treatment and Resolution of Venous Stasis Leg Ulcers
Brief Title: The Effects of Pulsed Elelectro-Magnetic Fields ("PEMF") in the Treatment of Venous Stasis Leg Ulcers
Acronym: VSLU
Status: Terminated | Type: Observational
Why Stopped: Dr. Siddiqui, the principal investigator, was unable to continue recruiting during and after covid.
Sponsor: PEMF Systems, Inc. (Industry)
Collaborators: Henry Ford Health System (Other)
Responsible Party: Sponsor
Other Study IDs: PEMF 102
Record Dates: First submitted 2017-04-05; First posted 2018-01-30 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Venous Stasis Ulcers
Keywords: ulcers; leg ulcers; venous stasis; ulcer treatment; leg ulcer treatment; venous stasis treatment; non invasive treatment; pulsed electromagnetic; pulsed electromagnetic therapy; pulsed electromagnetic treatment; pulsed magnetic; pulsed magnetic therapy; pulsed magnetic treatment; varicose Ulcer; ulcer pain
MeSH Terms: conditions — Varicose Ulcer; Ulcer; Leg Ulcer | interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Ulcer fluid .5 ml and blood 5 ml samples will be obtained for the following tests:
  Transforming Growth Factor ("TGF") Vascular Endothelial Growth Factor ("VEGF") Matrix Metalloroteinase ("MMP"), MMP-9 and MMP-13 Tumor Necrosis Factor alpha ("TNFα") Pro-inflammatory Cytokines: IL-1 α /IL-1F1 and IL-6
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- High-power PEMF device: 20 participants with VSLU will receive PEMF therapy with a high-power PEMF device for 10 minutes twice a day for each VSLU area.
  Interventions: Device: PEMF therapy with a high-power PEMF device
- Medium-power PEMF device: 20 participants with VSLU will receive PEMF therapy with a medium-power PEMF device for 15 minutes twice a day per VSLU area.
  Interventions: Device: PEMF therapy with a medium PEMF power device
- Low-power PEMF device: 20 participants with VSLU will receive PEMF therapy with a low-power PEMF device for 30 minutes twice a day per VSLU area..
  Interventions: Device: PEMF therapy with a low-power PEMF device
- Sham PEMF device: 20 participants with VSLU will receive PEMF therapy with a sham PEMF device identical to the low-power PEMF device and will treat each VSLU area for 15 minutes twice a day.
  Interventions: Device: PEMF therapy with the sham PEMF device

INTERVENTIONS:
Device: PEMF therapy with a high-power PEMF device — The 20 participants assigned to a high-power PEMF device will treat each Venous Stasis Leg Ulcer (VSLU) area for 10 minutes twice a day.
  Other Names: PEMF therapy with the Regenetron Pro; A; B; C; D
  Groups: High-power PEMF device
Device: PEMF therapy with a medium PEMF power device — The 20 participants assigned to a medium-power PEMF device will treat each VSLU area for 15 minutes twice a day.
  Other Names: PEMF therapy with the Regenetron Plus; A; B; C; D
  Groups: Medium-power PEMF device
Device: PEMF therapy with a low-power PEMF device — The 20 participants assigned to a low-power PEMF device will treat each VSLU area for 30 minutes twice a day.
  Other Names: PEMF therapy with the Regenetron; A; B; C; D
  Groups: Low-power PEMF device
Device: PEMF therapy with the sham PEMF device — The 20 participants assigned to the sham PEMF device will treat each VSLU area for 15 minutes twice a day.
  Other Names: PEMF therapy with the Regenetron sham; A; B; C; D
  Groups: Sham PEMF device

SUMMARY:
The purpose of this study is to determine the clinical effectiveness of a low-power PEMF device, a medium-power PEMF device and a high-power PEMF device as compared to a sham device to treat leg ulcers resulting from venous stasis ("VSLU").

DETAILED DESCRIPTION:
This study will demonstrate whether PEMF therapy is an effective adjunct treatment to the traditional treatment protocol used for the resolution of VSLU and of the pain associated with them. This is a 4 arm study done by comparing the outcomes of treatment with a low-power PEMF device, a medium-power PEMF device and a high-power PEMF device against those obtained from the control group treated with a sham PEMF device.

A device usability study is included in the study protocol to evaluate the participants' understanding of the device packaging, the User Manual, the device labeling, the controls and the directions for use. An un-blinded assistant ("UA") will manage the device usability study and hand out all informational literature and instructions to each participant, in accordance with the randomization protocol. Participants' success will be rated and their perception on the ease of use and how to make the device easier to use will be solicited.

Safety precautions and contraindications are specifically defined, and adverse/ unexpected events and reactions, if any, will be documented as they arise.

The primary aims of the study are to assess the effects of 16 weeks of PEMF treatment on the VSLU with one of three PEMF devices of different power levels against a sham PEMF device. The study has 3 specific aims:

Aim 1 (Primary) Determine if the use of specific PEMFs affect the time for healing trajectory of VSLU. Healing trajectory over the 16 week of the study protocol will be measured as the area under the curve for total lesion area expressed as a percentage of the baseline area.

Aim 2 (Secondary) Determine if VSLU and serum levels of three inflammatory cytokines: IL-1, IL-6 and TNF-alpha are affected by the use of specific PEMFs.

Aim 3 (Secondary) Determine if VSLU pain is improved by the use of specific PEMFs. Pain levels will be assessed with the use of allowed pain medication use by each participant. Pain will also be assessed with the five (5) pain scales from the National Initiative on Pain Control pain assessment scales ("NIPC scales") that will help each participant describe his/her pain levels and characteristics both quantitatively and qualitatively.

Eighty participants will be enrolled on the basis of leg ulcers due to venous insufficiency (VSLU) alone unless there are exclusions factors. The 80 participants will be divided in four groups of 20 participants: three treatment groups and a control group. Of the initial 80 participants at the investigation site approved to participate in this study, the outcome data of a net total of 72 participants, 18 per group, will be considered for analysis. The randomization protocol used for this study will occur in two stages: first with the blinding of the participants and the random assignment of a unique record number ("URN") to each of them and, second, with the random allocation of one of the PEMF or sham devices to each participant. Device allocation will be done according to a computer-generated table of random permutations designed to balance the number of participants in each group. All the data from the follow-ups, various assessments and testing procedures will be collected under the study URN for each participant. The URNs will be kept in a URN Record Log and kept in a locked cabinet in the principal investigator ("PI") 's office. Aside from the UA who will not be involved in data collection, monitoring or analysis, the investigators will be blinded to the URN assignment and to the PEMF or sham treatment protocol followed by each participant during the study. The randomization will not be broken until all eighty participants have completed the study.

The required effect sizes are all large; however, the PEMF effects are expected to be very large. The sample size of 80 participants provides required large effect sizes. Twenty patients will be enrolled per group and 18 are expected to have enough data to be included in the analysis.

Aim 1 With 20 participants enrolled in each of four arms, and a net sample size of 18 per group (accounting for 10% with incomplete data) and a p-value of 0.017 required for significance, there will be 80% power for a t-test to detect an effect size of 1.1 (i.e. a difference in mean area under the curve equal to 1.1 standard deviations). The secondary analysis for time to complete healing will have 80% power to detect a hazard ratio of 3.0.

Aim 2 and 3 The power for the multivariate test will be approximated by that available for a two sample t-test. With a net sample size of 18 per group and a p-value of 0.017 required for significance, the effect size will need to be 1.1 in order to have 80% power for a t-test. For the Wilcoxon rank sum test, the effect size may be expressed by the quantity Prob(X < Y) where X and Y are drug usage values from a random control group patient and a random patient from one of the PEMF groups. Under the null hypothesis, Prob(X < Y) = 0.5. With a sample size of 18 per group and alpha = 0.017, there will be 80% power to detect Prob(X < Y) = 0.81.

The Project Director, a direct agent of the company sponsoring the study, will periodically visit the research site to ensure the study is conducted in compliance with the approved Clinical Investigation Protocol and that the PI, the research assistant ("RA") and the UA adhere to the Protocol.

A record of the number of all screened participants, participants who refuse entry, and those entered in the study will be kept by the UA to follow CONSORT guidelines. He or she will also be informed and keep a record of any dropouts and the reason the participant was dropped from the study.

Statistical data will include 2 series of survey questionnaires at baseline and at the end of the study. The questionnaires include: Your Health in General (SF-36) and pain assessment using the National Initiative on Pain Control pain ("NIPC") assessment scales. A count, measurement and imaging of the VSLU using Silhouette High Tech cameras. Pain levels and pain medication intake will also be obtained weekly using a Caregiver Diary. A fluid and a small blood sample will be collected weekly from the VSLU area and tested for various inflammation biomarkers and growth factors. The data will be noted using a series of case report forms.

The primary tests for a PEMF benefit will be made using a Hochberg adjustment to take into account testing a single primary outcome measure (healing trajectory) measured three times, once for each of three different PEMF variations versus control. Under the Hochberg method, if all three primary test p-values are under 0.05, then all three will be considered significant. However, if only one is under 0.05, it will need to be under 0.05/3 = 0.017 in order to be considered significant. Assuming at least one of the PEMF variations is superior to control for at least one of the outcomes, a secondary analysis will compare each of the PEMF variations to the other two. A Hochberg adjustment will also be made for each of the two sets of secondary comparisons (pain and cytokines).

Aim 1 (Primary) The healing trajectory over 16 weeks will be compared for each PEMF variation versus the control group by t-test. Healing trajectory will be measured as the area under the curve for total lesion area expressed as a percentage of the baseline area.

Secondary analysis will use a log rank test to compare the times to complete healing. Descriptive analysis will plot the number of ulcers and their combined area over time for each subject. Kaplan-Meier survival curves for the time to complete healing will also be produced.

Aim 2 (Secondary) A multivariate test will be made comparing each PEMF group versus control, for a vector made up of the three cytokines: IL-1, IL-6 and TNF-alpha.

Aim 3 (Secondary) A multivariate test will be made comparing each PEMF group versus control, for a vector made up of the five pain scales. Pain medication usage will also be summarized using two quantities: a morphine equivalent dose to summarize all opioid drugs used, and a maximum dose equivalent for NSAIDs. Averages for these two medication use measures will be computed for the 16 weeks of observations and each will be analyzed separately using a Wilcoxon rank sum test.

The blinding assessment will occur at the end of the treatment protocol. Participants and investigators will be probed as to the device and treatment protocol each received.

All data, resulting analyses, and reports will remain proprietary to the sponsor. All case report forms and final data reports will be submitted to the sponsor for review and approval prior to any publication being made.

The data obtained from this study will demonstrate whether treatment with specific PEMFs affect the time for healing trajectory of VSLU; affect VSLU and serum levels of inflammatory cytokines; and if VSLU pain is improved.

A successful resolution of leg ulcers from venous stasis and the associated pain using therapeutic means, such as PEMF therapy, that are conservative, non-invasive, non-pharmacological and with no known undesirable side effects may prove to be quite significant.

ELIGIBILITY:
Inclusion Criteria:

Participants must also have normal cognitive and communicative abilities to provide comprehensive information for:

1. Health history questionnaire and Your Health in General ("SF-36")
2. The National Initiative on Pain Control pain assessment scales (NIPC scales). The NIPC scales are comprised of four complementary pain assessment rating scales, the Wong-Baker FACES Pain Rating Scale, Numeric Rating Scale (NRS), a pain location chart and a Pain Quality Assessment Scale© (PQAS©)

Exclusion Criteria:

1. Inability to obtain informed consent from participant
2. Prisoners or convicts
3. Hemorrhagic tendencies, Purpura, hemophilia, or any cardiovascular diseases
4. Severe anemia, Hemoglobin < 8.5
5. Severe hypoalbumenemia, serum albumen , 2.6
6. Poorly controlled diabetes, A1cHgb > 12
7. Severe renal failure - serum creatinine > 2.5 or hemodialysis
8. Severe hepatic insufficiency: know cirrhosis, any degree of ascites, serum transaminases more than 3 times the upper limit of normal
9. Pregnancy - women of childbearing potential must agree to use adequate contraception during the study
10. HIV infection unless on retroviral therapy and viral load undetectable by PCR
11. Severe hypoxemia - chronic oxygen or ventilator therapy
12. Known cryoglobulinemia
13. Systemic antibiotic therapy for any indication within 5 days of screening
14. A fracture to the lower extremities in the last 6 weeks
15. Within 24 hours of any surgery or 2 weeks of surgery on internal organs
16. Critically ill patients, patients hospitalized and patients who received transplants in past 2 months or patients in whom over-medication may be contraindicated
17. Active chemotherapy, cancer or malignant tumors
18. Any metal screws, pins and/or metallic implants within 15 inches of the VSLU
19. Participants with specific ulcers originating from sickle cell anemia or clinically significant infections as determined by ulcer culture
20. A history of difficult venipuncture for obtaining blood specimens
21. Current use of systemic agents or immunosuppressive therapy that may influence wound healing, such as Prednisone, Dexamethasone. Topical steroids to a maximum level of 25 mg Hydrocortisone daily applied no closer than 2.5 cm from the VSLU margin. Non steroidal anti-inflammatory drugs (NSAIDs) are not allowed except Ibuprofen maximum daily dose of 1800 mg, Acetaminophen maximum daily dose of 2600 mg (with or w/o opiates) and Naproxen maximum daily dose of 1000 mg
22. Current participation in any other clinical trial or study
23. Current involvement in a medical litigation or malpractice lawsuit.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participant population to be selected and studied will include male and female patients of all ethnic backgrounds ages 21 and older with one or more venous stasis leg ulcers (VSLU).
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Specific pulsed electromagnetic fields improves the healing trajectory of venous stasis ulcers. | The data necessary to establish the healing trajectory is collected over 16 weeks
  The healing trajectory will be evaluated after 16 weeks of PEMF treatment with one of three PEMF devices of different power level or a sham device. Leg ulcer area will be documented and a healing timeline will be defined. If healing is complete prior to the end of the 16-week treatment protocol, the RA will compile the length of time required for healing.

SECONDARY OUTCOMES:
Blood and serum levels of three inflammatory cytokines are affected by the use of specific pulsed electromagnetic fields. | The blood and serum samples are collected over 16 weeks
  The assessments will be evaluated after 16 weeks of PEMF treatment with one of three PEMF devices of different power level or a sham device. A fluid sample will be taken from the ulcer and a blood sample will be obtained from the participant. Both samples will be spun and placed at -70 degrees C. Serum and blood analyses will include a cytokine panel with IL-1, IL-6 and TNF-α. The following biomarkers: Transforming Growth Factor ("TGF") , Vascular Endothelial Growth Factor ("VEGF"), pro-inflammatory cytokines including IL-1 and IL-6, and Matrix Metalloroteinase ("MMP"), MMP-9 and MMP-13 will also be compared.
  The study will be terminated for each participant upon the healing of the venous leg ulcer(s) or at 16 weeks upon completion of the study, whichever comes first.
Venous leg ulcer pain is affected by the use of specific pulsed electromagnetic fields. | The assessments are collected over 16 weeks
  Pain levels will be recorded weekly and evaluated after 16 weeks of PEMF treatment within one of three PEMF devices of different power level or a sham device. Pain medication intake records from a Caregiver Diary and weekly follow-up medical examinations that will include an evaluation of pain using the National Initiative on Pain Control pain assessment scales (NIPC scales) will be collected and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Siddiqui, MD, Principal Investigator — Division Head, Plastic Surgery, Henry Ford Hospital; Guillemette Epailly, BS, MArch, Study Director — PEMF Systems, Inc.
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strauch B, Herman C, Dabb R, Ignarro LJ, Pilla AA. Evidence-based use of pulsed electromagnetic field therapy in clinical plastic surgery. Aesthet Surg J. 2009 Mar-Apr;29(2):135-43. doi: 10.1016/j.asj.2009.02.001. PMID 19371845
- [Background] Rohde C, Chiang A, Adipoju O, Casper D, Pilla AA. Effects of pulsed electromagnetic fields on interleukin-1 beta and postoperative pain: a double-blind, placebo-controlled, pilot study in breast reduction patients. Plast Reconstr Surg. 2010 Jun;125(6):1620-1629. doi: 10.1097/PRS.0b013e3181c9f6d3. PMID 20527063
- [Background] Stiller MJ, Pak GH, Shupack JL, Thaler S, Kenny C, Jondreau L. A portable pulsed electromagnetic field (PEMF) device to enhance healing of recalcitrant venous ulcers: a double-blind, placebo-controlled clinical trial. Br J Dermatol. 1992 Aug;127(2):147-54. doi: 10.1111/j.1365-2133.1992.tb08047.x. PMID 1390143
- [Background] Duran V, Zamurovic A, Stojanovic S, Poljacki M, Jovanovic M, Durisic S. [Therapy of venous ulcers using pulsating electromagnetic fields--personal results]. Med Pregl. 1991;44(11-12):485-8. Croatian. PMID 1821449
- [Background] Athanasiou A, Karkambounas S, Batistatou A, Lykoudis E, Katsaraki A, Kartsiouni T, Papalois A, Evangelou A. The effect of pulsed electromagnetic fields on secondary skin wound healing: an experimental study. Bioelectromagnetics. 2007 Jul;28(5):362-8. doi: 10.1002/bem.20303. PMID 17486634
- [Background] Itoh M, Montemayor JS Jr, Matsumoto E, Eason A, Lee MH, Folk FS. Accelerated wound healing of pressure ulcers by pulsed high peak power electromagnetic energy (Diapulse). Decubitus. 1991 Feb;4(1):24-5, 29-34. PMID 1994961
- [Background] Ieran M, Zaffuto S, Bagnacani M, Annovi M, Moratti A, Cadossi R. Effect of low frequency pulsing electromagnetic fields on skin ulcers of venous origin in humans: a double-blind study. J Orthop Res. 1990 Mar;8(2):276-82. doi: 10.1002/jor.1100080217. PMID 2303961
- [Background] Alekseenko AV, Gusak VV. [Treatment of trophic ulcers of the lower extremities using a magnetic field]. Klin Khir (1962). 1991;(7):60-3. Russian. PMID 1942838
- [Result] Kuliev RA, Babaev RF. [A magnetic field in the combined treatment of suppurative wounds in diabetes mellitus]. Vestn Khir Im I I Grek. 1992 Jan;148(1):33-6. Russian. PMID 1338829
- [Result] Alekseenko AV, Gusak VV, Stoliar VF, Iftodii AG, Tarabanchuk VV, Shcherban NG, Naumets AA. [Use of magnetic therapy combined with galvanization and tissue electrophoresis in the treatment of trophic ulcers]. Klin Khir (1962). 1993;(7-8):31-4. Russian. PMID 8139189
- [Result] Comorosan S, Vasilco R, Arghiropol M, Paslaru L, Jieanu V, Stelea S. The effect of diapulse therapy on the healing of decubitus ulcer. Rom J Physiol. 1993 Jan-Jun;30(1-2):41-5. PMID 7982015